CLINICAL TRIAL: NCT05241704
Title: Endovenous Ablation of Superficial Venous Reflux Combined With Fat Grafting Vs Endovenous Ablation Alone for the Treatment of Patients With Venous Ulcers: A Prospective Randomised Clinical Pilot Study
Brief Title: Endovenous Ablation Combined With Fat Grafting for Venous Ulcers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University of Ireland, Galway, Ireland (Other)
Responsible Party: Principal Investigator, Mohamed Elsharkawi, Principal Investigator, National University of Ireland, Galway, Ireland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 117/12
Record Dates: First submitted 2022-01-24; First posted 2022-02-16 (Actual); Last update posted 2022-02-16 (Actual); Status verified 2022-02

CONDITIONS: Varicose Ulcer
Keywords: venous, ulcers, fat graft, adipose, stem cells
MeSH Terms: conditions — Varicose Ulcer; Ulcer

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endovenous ablation of superficial venous reflux + Fat grafting (Experimental): Endovenous ablation of the main truncal venous reflux to the lowest point of incompetence, where possible (routine practice) + Fat grafting
  Interventions: Procedure: Fat grafting; Procedure: Endovenous ablation of superficial venous reflux
- Endovenous ablation of superficial venous reflux only (Active Comparator): Endovenous ablation of the main truncal venous reflux to the lowest point of incompetence, where possible (routine practice)
  Interventions: Procedure: Endovenous ablation of superficial venous reflux

INTERVENTIONS:
Procedure: Fat grafting — Under general or local anaesthesia, fat will be harvested from either abdomen or lower limb. After harvesting the fat by liposuction, the lipoaspirate will be injected underneath the ulcer under complete aseptic operative setting
  Arms: Endovenous ablation of superficial venous reflux + Fat grafting
Procedure: Endovenous ablation of superficial venous reflux — Endovenous ablation of the main truncal venous reflux to the lowest point of incompetence, where possible (routine practice)

SUMMARY:
The aim of this trial is to determine if fat grafting may have applicability to venous ulcers by comparing healing and recurrence rates in patients who receive combined fat grafting and endovenous ablation with patients who receive endovenous ablation only

DETAILED DESCRIPTION:
Study design:

This is a randomised, prospective, active-control pilot study to compare the effectiveness of fat grafting combined with endovenous ablation to endovenous ablation alone on wound healing in patients with venous ulcers in a tertiary vascular care centre. This study will randomise 20 patients with venous ulcers in an equal ratio to one of two treatment arms. The intervention arm will be randomised to undergo endovenous ablation of superficial venous reflux combined with fat grafting at the same setting. The control arm will be offered endovenous ablation only. All patients in both arms will receive compression therapy until full ulcer healing. They will then be followed up in the outpatient clinic every 4 weeks to record wound size and to monitor any adverse events.

Study setting:

Potential participants will be identified, screened and randomised at the vascular outpatient clinics within the Saolta group university hospitals, Ireland. Patients in both arms will receive the intervention in operating theatre in Roscommon University Hospital (RUH). Fat grafting will be performed under the supervision of a plastic surgeon. The coordinating centre will be the Department of Vascular and Endovascular Surgery, University College Hospital Galway (UCHG), and the School of Medicine at the National University of Ireland Galway (NUI Galway).

Study screening:

Patients with chronic venous ulcers will be invited to join the study. Researchers will screen the patient for inclusion and exclusion criteria. Invited patients will be provided with a pre-designed information leaflet. This leaflet will be fully explained to the patient at the initial assessment. The study researchers will answer any questions about the study. Informed consent will be obtained from the patient on a formatted consent form. Patients will be given the freedom to give consent either on the same day or later.

Baseline visit:

Patients will undergo detailed clinical assessment by the researcher as part of the baseline evaluation. Recorded assessments will include:

* Demographics
* General clinical details (ABPI, comorbidities, medication history)
* Ulcer details (location, duration, size, progression, previous ulcer history). If the patient has multiple venous ulcers, we will only report on the largest of these ulcers as the index ulcer.
* Details of venous disease (previous deep vein thrombosis, previous venous interventions, pattern of venous reflux on duplex)
* Assessment of Clinical, Etiologic, Anatomic, Pathophysiological (CEAP) score via performing venous duplex scan.
* Disease specific and quality of life assessment scores

Sample size:

There are currently no previous studies from which we can withdraw a power calculation for this trial. Previous studies on the use of fat grafting have looked at fat grafting as a sole intervention. To our knowledge there are no studies that have combined both endovenous ablation and fat grafting. As such this study is designed as a pilot study. The proposed sample size for this pilot study is 20 patients, being randomised to 10 patients in each arm.

Randomisation:

After meeting the inclusion criteria, screened patients will be randomised to one of two treatment arms. The intervention arm will receive fat grafting combined with endovenous ablation. The control arm will be offered endovenous ablation only. This is an intention to treat designed study, where patients are analysed as randomised. Each screened patient will be given a unique screening number.

Sequence generation:

Screened patients will be randomised in a 1:1 ratio of study intervention: control according to a randomisation scheme. The randomisation scheme will be produced using the PROC PLAN® procedure of the SAS® software package (version 9.2.2) using a simple randomisation strategy. The scheme will be concealed from all patients and study personnel until after database lock.

Allocation concealment:

Patients will be allocated to intervention via a sequentially numbered opaque sealed envelopes, which will not deliver the randomised allocation except after registering the subject screening number. Each screened patient who is recruited to the trial will be given a unique patient trial number.

Blinding:

It will be impossible to blind the investigator and the patient due to the obvious difference in the surgical approach. Outcome assessors will be blinded. However, in the event of an adverse event outcome assessors will be unblinded.

Statistical analysis:

All data will be analysed according to the intention to treat principle. The comparison of the primary outcomes measure (time to healing) achievement in the two arms will be performed by using Kaplan Meier survival curves and Log rank test. Secondary outcomes will be assessed using Chi square or Fisher's Exact, where appropriate. An exact 95% confidence interval will be applied for the difference between intervention groups.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or more.
* Able to provide written informed consent.
* Chronic venous ulcers (C6 on CEAP classification).
* Superficial venous disease diagnosed on venous duplex.
* Ankle-brachial pressure index (ABPI) of 0.8 or more.

Exclusion Criteria:

* Evidence of deep venous occlusion
* Infected ulcers
* Malignancy or immune-suppression
* Malnutrition
* Multi-organ failure
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-02 (Estimated); Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Time to ulcer healing | 12 weeks
  Defined as time needed for complete re-epithelialisation with no dressing required post procedure

SECONDARY OUTCOMES:
Ulcer healing rates | 12 weeks
  Defined as proportion of ulcers fully healed at 12 weeks post procedure
Recurrence rates | 1 year
  Defined as proportion of new onset break down of epithelium in a fully healed index post procedure ulcer within 12 months post intervention
Incidence of adverse events | 1 year
  bleeding, infection, failure, thrombophlebitis, pulmonary embolism, nerve injury, fat embolism and fat necrosis
Visual Analog Score for pain | 1 year
  Visual Analog Score for pain, 0-10, 10 is the worst
The Aberdeen Varicose Vein Questionnaire (AVVQ) | 1 year
  from 0-100 (0 is the best possible quality of life and 100 the worst)
The quality of life score *EuroQol-5D (EQ-5D) | 1 year
  from 0-100 (0 is the worst possible health status and 100 is the best)
The quality of life score SF36 | 1 year
  The Short-Form (SF36), The lower the score the more disability

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Elsharkawi, Principal Investigator — University College Hospital Galway
Locations (1):
- Galway University Hospital, Galway, Ireland

IPD SHARING:
Plan to Share IPD: No